CLINICAL TRIAL: NCT01093235
Title: ARTemis - Avastin Randomized Trial With Neo-Adjuvant Chemotherapy for Patients With Early Breast Cancer
Brief Title: Combination Chemotherapy With or Without Bevacizumab in Treating Patients With Nonmetastatic Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000668530; CRCA-CCTC-WCTU-ARTemis; ISRCTN68502941; EUDRACT-2008-002322-11; EU-21017; MREC-08/H1102/104
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer; Cardiac Toxicity; Perioperative/Postoperative Complications
Keywords: cardiac toxicity; perioperative/postoperative complications; HER2-negative breast cancer; male breast cancer; estrogen receptor-negative breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-negative breast cancer; progesterone receptor-positive breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Postoperative Complications; Breast Neoplasms, Male; Inflammatory Breast Neoplasms | interventions — Bevacizumab; Cyclophosphamide; Docetaxel; Epirubicin; Fluorouracil; Neoadjuvant Therapy

INTERVENTIONS:
Biological: bevacizumab
Drug: cyclophosphamide
Drug: docetaxel
Drug: epirubicin hydrochloride
Drug: fluorouracil
Procedure: assessment of therapy complications
Procedure: neoadjuvant therapy
Procedure: quality-of-life assessment
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, fluorouracil, epirubicin hydrochloride, and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving combination chemotherapy together with or without bevacizumab is more effective in treating patients with nonmetastatic breast cancer.

PURPOSE: This randomized phase III trial is studying how well giving combination chemotherapy works compared with giving combination chemotherapy together with bevacizumab in treating patients with nonmetastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of neoadjuvant therapy comprising docetaxel, fluorouracil, epirubicin hydrochloride, and cyclophosphamide with versus without bevacizumab in patients with HER2-negative nonmetastatic breast cancer.

Secondary

* To assess quality of life of female patients treated with these regimens.

OUTLINE: This is a multicenter study. Patients are stratified according to age (≤ 50 years old vs > 50 years old), estrogen receptor status (negative [Allred score 0-2] vs weakly positive [Allred score 3-5] vs strongly positive [Allred score 6-8]), total tumor size* (≤ 50 mm vs > 50 mm), clinical involvement of axillary nodes (yes vs no), and inflammatory/locally advanced disease (T4) (yes vs no). Patients are randomized to 1 of 2 treatment arms.

NOTE: *In cases with multifocal disease in one breast, or bilateral disease, the size to be used for the stratification is the sum of the single largest diameter of all measurable tumors.

* Arm I: Patients receive docetaxel IV on day 1; treatment repeats every 3 weeks for 3 courses. Patients then receive fluorouracil IV, epirubicin hydrochloride IV, and cyclophosphamide IV on day 1 (FEC). Treatment with fluorouracil, epirubicin hydrochloride, and cyclophosphamide repeats every 3 weeks for 3 courses.
* Arm II: Patients receive bevacizumab IV over 30 to 90 minutes and docetaxel IV on day 1; treatment repeats every 3 weeks for 3 courses. Patients then receive FEC as in arm I. Treatment with FEC repeats every 3 weeks for 3 courses. Patients also receive bevacizumab IV over 30 to 90 minutes and docetaxel IV on day 1 in FEC course 1 only.

Within 3-6 weeks after completion of last dose of study therapy, patients in both arms undergo surgery. Within 4-8 weeks after surgery, patients undergo radiotherapy according to standard protocol.

Women complete quality-of-life questionnaires (FACT-B and EuroQoL) at baseline and during and after completion of study treatment.

After completion of study treatment, patients are followed every 6 months for 2 years and then annually for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer
* HER2-negative disease

  * IHC 0/1 OR IHC 2+ and FISH negative
* Must meet 1 of the following criteria:

  * Unifocal tumor meeting 1 of the following criteria:

    * T2 or T3 tumors (radiological size > 20 mm)
    * T4 tumor of any size with direct extension to the chest wall or the skin
    * Inflammatory carcinoma with tumor of any size
  * Multifocal tumor meeting the following criteria:

    * The sum of each tumors' maximum diameter must be ≥ 20 mm (total radiological tumor size ≥ 20 mm)
  * Other locally advanced disease meeting 1 of the following criteria:

    * Any T stage with involvement of large or fixed axillary lymph nodes (radiological diameter > 20 mm or clinical N2) and primary breast tumor of any diameter
    * Any T stage with involvement of large or fixed axillary lymph nodes (radiological diameter > 20 mm or clinical N2), without a primary breast tumor identified and the presence of breast cancer in a lymph node must be histopathologically confirmed by lymph node biopsy (tru-cut or whole lymph node)
* Embedded paraffin tumor block available from pre-chemotherapy biopsy and surgical specimen
* Bilateral disease allowed
* No evidence of metastatic disease
* No prior breast cancer except for ductal carcinoma in situ of the breast surgically cured > 10 years ago
* Any hormone receptor status

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC > 3 x 10^9/L
* Hemoglobin > 10 g/dL
* Platelet count > 100 x 10^9/L
* AST/ALT ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2 times ULN
* Bilirubin normal

  * Isolated elevation of bilirubin to ≤ 3 times ULN with a presumptive diagnosis of Gilbert syndrome allowed if AST/ALT and alkaline phosphatase are within normal limits
* Creatinine ≤ 1.5 times ULN
* PT and PTT/aPTT ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* Must be fit to receive chemotherapy on this trial, in the opinion of the responsible clinician, as indicated by the following criteria:

  * No clinically significant cardiac abnormalities
  * No myocardial infarction within the past 6 months
  * LVEF normal (at least 50%) by MUGA scan or echocardiogram
* No prior ischemic heart disease, cerebrovascular disease, peripheral vascular disease, arterial or venous thromboembolic disease, cardiac failure, inflammatory bowel disease, gastroduodenal ulcer, symptomatic diverticulitis, or bleeding diathesis
* No uncontrolled hypertension (systolic BP > 150 mm Hg or diastolic BP > 90 mm Hg) with or without antihypertensive medication

  * Patients with initial blood pressure elevations are eligible provided initiation or adjustment of antihypertensive medication lowers pressure to meet entry criteria
* No other previous malignancy except basal cell carcinoma, carcinoma in situ of the cervix, or ductal carcinoma in situ of the breast treated by surgery only and disease-free for 10 years
* No concurrent medical or psychiatric problem that might prevent completion of treatment or follow-up
* No presence of active uncontrolled infection
* No history of nephritic or nephrotic syndrome
* No traumatic injury within the past 28 days
* No evidence of other disease that, in the opinion of the investigator, places the patient at high risk of treatment-related complications
* No nonhealing wound, peptic ulcer, or bone fracture

PRIOR CONCURRENT THERAPY:

* No prior neoadjuvant endocrine therapy
* No prior chemotherapy or radiotherapy
* No major surgical procedure within the past 28 days
* No concurrent full therapeutic dose of anticoagulants or aspirin > 325 mg/day, clopidogrel > 75 mg/day, or corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Complete pathological response rates (tumor and lymph nodes)

SECONDARY OUTCOMES:
Disease-free survival
Overall survival
Pathological complete response rate in breast alone
Radiological response after 3 and 6 courses of chemotherapy
Rate of breast conservation
Toxicities, including cardiac safety and surgical complications (wound healing, bleeding, and thrombosis)
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Helena Earl, MBBS, PhD, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, England, United Kingdom

REFERENCES:
- [Derived] Ali HR, Dariush A, Thomas J, Provenzano E, Dunn J, Hiller L, Vallier AL, Abraham J, Piper T, Bartlett JMS, Cameron DA, Hayward L, Brenton JD, Pharoah PDP, Irwin MJ, Walton NA, Earl HM, Caldas C. Lymphocyte density determined by computational pathology validated as a predictor of response to neoadjuvant chemotherapy in breast cancer: secondary analysis of the ARTemis trial. Ann Oncol. 2017 Aug 1;28(8):1832-1835. doi: 10.1093/annonc/mdx266. PMID 28525534
- [Derived] Earl HM, Hiller L, Dunn JA, Blenkinsop C, Grybowicz L, Vallier AL, Gounaris I, Abraham JE, Hughes-Davies L, McAdam K, Chan S, Ahmad R, Hickish T, Rea D, Caldas C, Bartlett JMS, Cameron DA, Provenzano E, Thomas J, Hayward RL; ARTemis Investigators Group. Disease-free and overall survival at 3.5 years for neoadjuvant bevacizumab added to docetaxel followed by fluorouracil, epirubicin and cyclophosphamide, for women with HER2 negative early breast cancer: ARTemis Trial. Ann Oncol. 2017 Aug 1;28(8):1817-1824. doi: 10.1093/annonc/mdx173. PMID 28459938
- [Derived] Earl HM, Hiller L, Dunn JA, Blenkinsop C, Grybowicz L, Vallier AL, Abraham J, Thomas J, Provenzano E, Hughes-Davies L, Gounaris I, McAdam K, Chan S, Ahmad R, Hickish T, Houston S, Rea D, Bartlett J, Caldas C, Cameron DA, Hayward L; ARTemis Investigators. Efficacy of neoadjuvant bevacizumab added to docetaxel followed by fluorouracil, epirubicin, and cyclophosphamide, for women with HER2-negative early breast cancer (ARTemis): an open-label, randomised, phase 3 trial. Lancet Oncol. 2015 Jun;16(6):656-66. doi: 10.1016/S1470-2045(15)70137-3. Epub 2015 May 11. PMID 25975632